CLINICAL TRIAL: NCT00658918
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Clinical Trial Designed to Assess the Safety of Ciclesonide, Applied as a Nasal Spray at Three Dose Levels, 200µg, 100µg or 25µg Once Daily for Six Weeks, in the Treatment of Perennial Allergic Rhinitis (PAR) in Pediatric Patients 2-5 Years of Age.
Brief Title: To Assess the Safety of Ciclesonide, Applied as a Nasal Spray at Three Dose Levels, in the Treatment of Perennial Allergic Rhinitis in Pediatrics (BY9010/M1-405)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BY9010/M1-405
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: Rhinitis, Allergic, Perennial; Hay Fever
Keywords: Perennial Allergic Rhinitis; Ciclesonide; Hay Fever; PAR
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- 1 (Active Comparator): Ciclesonide 200µg
  Interventions: Drug: Ciclesonide nasal
- 2 (Active Comparator): Ciclesonide 100µg
  Interventions: Drug: Ciclesonide nasal
- 3 (Active Comparator): Ciclesonide 25µg
  Interventions: Drug: Ciclesonide nasal
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide nasal — safety of Ciclesonide (200µg, 100µg, 25µg)
  Arms: 1; 2; 3
Drug: Placebo — placebo
  Arms: 4

SUMMARY:
The primary objective of this study is to demonstrate the safety of three dose levels of ciclesonide administered as an intranasal spray for six weeks, 200µg, 100µg or 25µg, once daily, in pediatric patients (ages 2-5 years) with PAR. The secondary objective is to measure serum concentrations of ciclesonide and its active metabolite under steady state conditions at three time points corresponding to the presumed peak and trough exposure after six weeks of administration.

In addition, reflective (24-hour) total nasal symptom score (TNSS) over the six weeks of treatment at various timepoints and a physician assessment of nasal symptoms at endpoint were summarized.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 2 and 5 years, inclusive
2. General good health, and free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the trial
3. A demonstrated sensitivity to at least one allergen known to induce PAR through a standard prick skin test within one year of study start. A positive test is defined as a wheal diameter at least 3mm larger than the control wheal for th eprick test
4. Parent or legal guardian is capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent and comply with all study requirements (visits, record-keeping, etc.)
5. A history of PAR for a minimum of 3 months preceding the study screening visit (B0). The PAR must have been of sufficient severity to require treatment (either continuous or intermittent) in the past and in the investigators judgment is expected to continue to require treatment for the study duration.

Exclusion Criteria:

1. History of physical findings of nasal pathology, including nasal polyps (within the last 60 days) or other clinically significant respiratory tract malformations, recent nasal biopsy (within the last 60 days), nasal trauma, or surgery and atrophic rhinitis or rhinitis medicamentosa (within the last 60 days).
2. Participation in any investigational drug trial within the 30 days preceding the Screening Visit (B0) or at any time during the trial
3. A known hypersensitivity to any corticosteroid or any of the excipients in the formulation.
4. History of a respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, the common cold, acute or chronic sinusitis, flu, severe acute respiratory syndrome (SARS)] within the 14 days preceding the Screening Visit, or development of a respiratory infection during the Screening Visit (B0)
5. History of a positive test for HIV, hepatitis B or hepatitis C.
6. Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of b-agonists and any controller drugs (e.g. theophylline, leukotrienes, etc.) intermittent use of b-agonists is acceptable
7. Use of any prohibited concomitant medications within the prescribed (per protocol) withdrawal periods prior to the screening visit (B0) and during the entire screening period and treatment duration
8. Use of antibiotic therapy for acute conditions within 14 days prior to the Screening Visit (B0).
9. Initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the Screening Visit AND use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
10. Non-vaccinated exposure to, or infection with, chickenpox or measles within the 21 days preceding the Screening Visit (B0).
11. Exposure to systemic corticosteroids for any indication, chronic or intermittent (e.g.: contact dermatitis), during the past 2 months, or presence of an underlying condition that can reasonably be expected to require treatment with corticosteroids during the course of the study.
12. Use of topical corticosteroids in concentrations in excess of 1% hydrocortisone for dermatological conditions during the past 1 month, or presence of an underlying condition that can reasonably be expected to require treatment with such preparations during the course of the study.
13. Intraocular pressure at the screening visit (B0) of 21 mm Hg or greater or failed reading at the screening Visit (B0)
14. Glaucoma requiring treatment
15. Use of antiepileptic drugs for epilepsy within 30 days of the screening visit (B0) or anytime during the treatment period.
16. Initiation of pimecrolimus 1% cream or tacrolimus ointment 0.1% or 0.03% during the study period or planned dose escalation during the study period. However, initiation of these creams/ointments 30 days or more prior to the screening Visit (B0) AND use of a stable (maintenance) dose during the study period may be considered for inclusion

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2004-09; Primary Completion 2005-04 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Spontaneous and elicited adverse events (AEs) | 6 weeks
Vital signs | 6 weeks
Cortisol (24-hour urine. AM plasma) | 6 weeks
clinical laboratory parameters | 6 weeks
Physical examination including ENT exam | 6 weeks
Intraocular pressure (IOP) assessment | 6 weeks
serum concentrations of ciclesonide and its active metabolite will be measured following 6 weeks treatment at three time points corresponding to presumed peak and trough exposure | 6 weeks

SECONDARY OUTCOMES:
reflective (24-hour) total nasal symptom score (TNSS; including sneezing, runny nose, nasal itching and congestion) over 6 weeks of treatment and over other selected time points | 6 weeks
a physician assessment of nasal symptoms at endpoint and at Visits T0, T3 and T6 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Altana/Nycomed, Little Rock, Arkansas, United States

REFERENCES:
- See also: BY9010-M1-405-RDS-2005-11-07.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4533&filename=BY9010-M1-405-RDS-2005-11-07.pdf